CLINICAL TRIAL: NCT04271891
Title: the Effect of WBPC on Subacute Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Wei-Te Wang, Attending physician of physical medicine and rehabilitation, Changhua Christian Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCH_101101; 100-CCH-IRP-62
Record Dates: First submitted 2019-01-30; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- With WBPC (Experimental): Intensive rehabilitation programs :The duration will be 30 minutes a time, and the frequency will be 5 days a week, and the treating period will be 3 weeks additional WBPC: The duration will be 30 minutes a time
  Interventions: Device: WBPC
- Control (Placebo Comparator): Intensive rehabilitation programs: The duration will be 30 minutes a time, and the frequency will be 5 days a week, and the treating period will be 3 weeks without WBPC.
  Interventions: Device: Without WBPC

INTERVENTIONS:
Device: WBPC — The duration will be 30 minutes a time, and the frequency will be 5 days a week, and the treating period will be 3 weeks.
  Arms: With WBPC
Device: Without WBPC — Not treat with WBPC
  Arms: Control

SUMMARY:
Whole body periodic acceleration (WBPA) is a head-to-toe movement. The function WBPA works as adding pulses to the circulation. This motion increases shear stress to the endothelium, which stimulates increased release of endothelial-derived nitric oxide (eNO), prostaglandin E-2, tissue plasminogen activator (TPA) into the circulation, and these substances are cardioprotective and contribute to vasodilatation. The WBPA were not well studied than whole body vibration (WBV), a vertical rocking training machine, and most researches focused on cardioprotective effects. A study revealed the effect of Moderate-Intensity Exercise and Whole-Body Periodic Acceleration on Nitric Oxide release was the same. This instrument is quite safe and was applied to patients with varied diseases in previous study. No sound contraindication was mentioned till now.

Our hypothesis is assuming that the circulation of brain could improve after the intervention of WBPA, and stroke recovery and cadio-pulmonary function will improve subsequently.

DETAILED DESCRIPTION:
So the investigators will recruit subacute stroke patients as our subjects. The patient who is booked to our rehabilitation ward for further rehabilitation programs is eligible for our study. the investigators will recruit 30 patients, and randomize them to experimental and control group. This study is going to be single blinded, which the evaluator is blinded to the condition of the subjects. Whether experimental or control groups will received the same intensive rehabilitation programs (6 days a week). The experimental group will receive additional WBPA treatment. The duration will be 30 minutes a time, and the frequency will be 5 days a week, and the treating period will be 3 weeks. The evaluator will assess twice, before and after the experiment period. The measurements include: muscle power, brunnstrom stages, Barthel Index, functional independence measure (FIM), time up and go test, 6 minutes walk test, Fugl-Meyer Assessment, berg balance scale, cardio-pulmonary test. In addition, to confirm the immediate effect of WBPA over brain circulation, the investigators will choose 6 patients to received carotid ultrasonography before and immediately after the WBPA treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subacute stroke patient onset 1-3 months, age from 40-80 years-old

Exclusion Criteria:

* Cognition impaired(MMSE<24), not first-ever stroke, MI history, AF, CHF, NIHSS>12

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Functional independent measurement(FIM) | up to 3 weeks
  Score from 18 to 126, assessment of degree of disability depends , 18 categories(score from 1~7 points, 1 = <25% independence; total assistance required, 7 = 100% independence), focusing on motor and cognitive function, Represent post-stroke patient's ADL function
Brunnstrom stage, | up to 3 weeks
  Stage I to V, stage I: flaccid ; stage II: spasticity appeared, associated movement; stage III: increased spasticity, synnergy movement; stage IV: decreased spasticity, breaking synergy; stgae V:most independent movement; stage VI: normal. Represent post stroke limb function
modified Ashworth Scale, | up to 3 weeks
  From 0 to 4 , evaluate post stroke patient's spasticity, 0: No increase in muscle tone; 1: Slight increase in muscle tone;1+: Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM; 2: More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved 3: Considerable increase in muscle tone, passive movement difficult;4: Affected part(s) rigid in flexion or extension

SECONDARY OUTCOMES:
quality of life: short form- 36 | up to 3 weeks
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability

CONTACTS AND LOCATIONS:
Locations (1):
- Changhua Christian Hospital, Changhua, Taiwan